CLINICAL TRIAL: NCT06297473
Title: Physical Attendance Versus Telephone or Video Follow-up for Prevention of Severe Adverse Events in Patients With Non-functioning Pituitary Tumors. A Pragmatic Randomized Controlled Multi-center Non-inferiority Trial.
Brief Title: Physical Attendance Versus Telephone or Video Follow-up in Patients With Non-functioning Pituitary Tumors.
Acronym: PITCARE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SJ-1050
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Functional Pituitary Adenoma

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either intervention or control
Who Masked: Outcomes Assessor
Masking Description: Adverse events (primary outcome) will be established by a blinded adjudication committee.
  A committé of external endocrinologist/ophthalmologist will blinded to participant ID/allocation assess all the participants admissions to hospital and assess wether it qualifies as an event
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone-/video follow-up (Experimental): Yearly routine review of patients status will take place by using telephone- or video consultation.
  Interventions: Behavioral: Telephone-/video follow-up
- Standard (Active Comparator): Yearly routine review of patients status will take place as an in-person interview
  Interventions: Behavioral: In-person follow-up

INTERVENTIONS:
Behavioral: Telephone-/video follow-up — The yearly routine review of patients takes place by using a telephone or video interview rather than in-person interview in the endocrine outpatient department.
  All other assessments, e.g. biochemical, MRI, is conducted as usual.
  Arms: Telephone-/video follow-up
Behavioral: In-person follow-up — The yearly routine review on patients takes place at the endocrine outpatient department
  Arms: Standard

SUMMARY:
The primary purpose of this study is to compare the safety of routine telephone assessment versus in-person assessment during a two-year period for patients with non-functioning pituitary adenomas. Secondly, to compare the quality of pituitary care in persons having biochemical assessment once versus twice a year. Thirdly, to assess the rationale of repeated assessment of pituitary function and imaging in patients with small pituitary tumors (microadenomas).

DETAILED DESCRIPTION:
This study intends to investigate the treatment quality, treatment safety, and patient satisfaction of increased use of telephone/video clinics compared to physical attendance during a three year period. Secondly, the study will assess the impact of reducing biochemical assessment by 50 % and explore the possibility of reducing patients with non-functioning pituitary tumors (NFPTs) affiliated to endocrine departments by 10 - 20 %.

Objective

1. The primary objective is to compare a phone/video follow-up versus standard follow-up in adults with stable non-functioning pituitary tumors for the risk of admission for acute adrenal crisis, poor visual outcome after pituitary surgery, or admission with hypo- or hypernatremia caused by diabetes insipidus.
2. Main secondary objective is to compare yearly endocrine check-up versus endocrine check-up every 6 months in adults with stable non-functioning pituitary tumors for adequate control of hormonal replacement therapy.
3. To assess whether hormonal replacement therapy in patients followed by phone/video consultation is non-inferior to patients followed with standard treatment.
4. Another secondary objective is to use the collected data to quantify the risk of surgery/radiotherapy of pituitary tumor due to tumor growth or new endocrinopathies in patients with micro-NFPTs.

Design This study is an investigator initiated pragmatic multicenter non-inferiority trial with blinded outcome assessment.

Trial procedure Eligible patients will be approached at the yearly routine visit for information of the trial. Patients fulfilling the inclusion criteria and none of exclusion criteria will offered enrollment in the trial. Patients will be randomized to either at standard treatment, planned yearly in-person visits for the next two years, or the intervention which is planned yearly control by telephone or video contact for the next two years. Following randomization there a no restrictions on patient care. Primary outcome will be assessed from randomization to the last visit (2 years from randomization) by a blinded adjudication committee.

A nurse or medical student will continuously monitor patient files for events. The study is planned to run from April 1st 2024 to January 1st 2028.

Information from patient files Once patients have accepted participation in the trial, information regarding previous disease history will be extracted. This include information on co-morbidity, development of pituitary MRI findings, development in ophthalmological findings, biochemistry, treatment related to pituitary failure, and treatment related to pituitary adenoma in the form of surgery or radiotherapy.

Intervention Participants allocated to the intervention-group will receive their annual endocrine review as a telephone or video contact for two years in a row. There will be no differences in endocrine review, e.g. biochemical assessment or MRI. Patients or treating physician can choose to make in-person assessment or follow-up if needed.

Comparator group Participants allocated to the comparator group will receive standard treatment with yearly in-person assessment, e.g. biochemical and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Non-functioning pituitary tumor
* Diagnosed > 6 months from enrollment, i.e. found on MRI.

Exclusion Criteria:

* Planned pituitary surgery
* Planned radiotherapy
* Poor Danish skills
* Patient is considered by the treating physician unsuitable for follow-up by telephone or video

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of adverse events | Two year period. From allocation including the routine follow-up after two years.
  The primary outcome is a composite outcome comprised of the three individual outcomes considered of equal importance to patients and clinicians: Risk of admission for adrenal crisis, risk of admission for severe hypo- or hypernatremia, risk of pituitary surgery with lack of full recovery of vision after surgery.

SECONDARY OUTCOMES:
Thyroid replacement therapy | At two years follow-up
  In patients on thyroid replacement therapy: Comparing levels of free T4.
Growth hormone replacement therapy | At two years follow-up
  In patients on growth hormone replacement therapy: Comparing IGF-1 levels
Desmopressin replacement therapy | At two years follow-up
  In patients on vasopressin replacement therapy: Comparing levels of sodium
Hormonal replacement therapy | At two years follow-up
  In patients on hormonal replacement therapy: Comparing levels of total testosterone in men and estradiol in women

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Krogh, DMSc, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
No current plan. If relevant researchers with relevant project plan approaches we are willing to share anonymous IPD.